CLINICAL TRIAL: NCT01336946
Title: Effectiveness and Cost-effectiveness of a Health Promotion Intervention Targeting Physical Activity and Eating Habits in Persons With Mental Disorders
Brief Title: HEalth Promotion Intervention in MEntal Health Care
Acronym: HEPIMEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC/2010/607
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Unhealthy Lifestyle of Persons With Mental Disorders
Keywords: lifestyle; mental disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- health promotion program (Experimental): Psycho education and behavioural group sessions and supervised walking sessions will be performed.
  Interventions: Behavioral: Psycho educational and behavioural group sessions; Behavioral: Walking session
- Control group (No Intervention): No intervention will be performed in this control group.

INTERVENTIONS:
Behavioral: Psycho educational and behavioural group sessions — 10 psycho educational and behavioural group sessions on topics like the Food Triangle, healthy eating, the importance of physical activity, healthy eating on a limited budget, implementing physical activity into the daily life, the influence of advertisements...
  Arms: health promotion program
Behavioral: Walking session — A weekly supervised walking session (30 minutes) in a 10-week period.
  Arms: health promotion program

SUMMARY:
Overweight and obesity have become a serious global public health problem and the prevalence of these conditions is even higher among persons with mental disorders, compared with the general population. Overweight and obesity are partially associated with sedentary lifestyles and unhealthy eating habits.

The aim of the study is to examine the effectiveness and cost-effectiveness of a health promotion intervention targeting physical activity and eating habits in persons with mental disorders.

The study hypothesis is that between baseline and the end of the intervention, and after a 6-month follow up period, significant differences in the primary and secondary outcomes between the intervention and control group will be identified. The investigators also hypothesize that the health promotion intervention will be cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* living in sheltered housing
* diagnosed according to the Diagnostic and Statistical Manual of mental disorders (DSM-IV manual)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change in body weight 10 weeks post-intervention | after 10 weeks
  The primary outcome of the study consists of changes in body weight between baseline and 10-weeks post-intervention in the intervention and control group separately and between the intervention and the control group.The participants will be weighed in light clothing without shoes, with standardised measurement.
change in body weight 26 weeks post-intervention | after 26 weeks
  The primary outcome of the study consists of changes in body weight between baseline and 26-weeks post-intervention in the intervention and control group separately and between the intervention and the control group.The participants will be weighed in light clothing without shoes, with standardised measurement.

SECONDARY OUTCOMES:
Body Mass Index 10 weeks post-intervention | after 10 weeks
  Body Mass Index, calculated as the weight in kilograms divided by the square of the height in metres (kg/m²)
Body Mass Index, 26 weeks post-intervention | after 26 weeks
  Body Mass Index, calculated as the weight in kilograms divided by the square of the height in metres (kg/m²).
Waist circumference, 10 weeks post-intervention | After 10 weeks
  Waist circumference, assessed by using a tape measure.
Waist circumference, 26 weeks post-intervention | After 26 weeks
  Waist circumference, assessed by using a tape measure.
Quality of Life, 10 weeks post-intervention | After 10 weeks
  Quality of life, assessed by using the SF-36 Health Survey.
Quality of Life, 26 weeks post-intervention | After 26 weeks
  Quality of life, assessed by using the SF-36 Health Survey.
Levels of physical activity, 10 weeks post-intervention | After 10 weeks
  Levels of physical activity, assessed by using the International Physical Activity Questionnaire long version (IPAQ) and by using pedometers.
Levels of physical activity, 26 weeks post-intervention | After 26 weeks
  Levels of physical activity, assessed by using the International Physical Activity Questionnaire long version (IPAQ) and by using pedometers.
Eating habits, 10 weeks post-intervention | After 10 weeks
  Eating habits, assessed by using a 24-hour dietary recall.
Eating habits, 26 weeks post-intervention | After 26 weeks
  Eating habits, assessed by using a 24-hour dietary recall.
Psychiatric symptom severity, 10 weeks post-intervention | After 10 weeks
  Psychiatric symptom severity, assessed by using the Brief Symptom Inventory (BSI).
Psychiatric symptom severity, 26 weeks post-intervention | After 26 weeks
  Psychiatric symptom severity, assessed by using the Brief Symptom Inventory (BSI).

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Annemans, Ph.D., Professor, Principal Investigator — University Ghent
Locations (25):
- Belgium (25):
  - Beschut Wonen Antwerpen, Antwerp
  - Beschut Wonen Min, Antwerp
  - Beschut Wonen Beernem, Beernem
  - Beschut Wonen De Raster, Beigem
  - Beschut Wonen Oostkust, Blankenberge
  - Beschut Wonen Brugge, Bruges
  - Beschut Wonen De Linde, Diest
  - Beschut Wonen De Wende, Eeklo
  - Beschut Wonen Centrum Onderweg, Ghent
  - Beschut Wonen Delta Wonen, Ghent
  - Beschut Wonen Domos, Ghent
  - Beschut Wonen Zagan, Ghent
  - Beschut Wonen Basis, Hasselt
  - Beschut Wonen West-Limburg, Heusden-Zolder
  - Beschut Wonen regio Izegem, Izegem
  - Beschut Wonen De Bolster, Kortrijk
  - Beschut Wonen De Hulster, Leuven
  - Beschut Wonen Het Veer, Maasmechelen
  - Beschut Wonen Eigen Woonst, Menen
  - Beschut Wonen Oostende, Ostend
  - Beschut Wonen Noord-Limburg, Overpelt
  - Beschut Wonen Roeselare-Tielt, Roeselare
  - Beschut Wonen Pro Mente, Sint-Niklaas
  - Beschut Wonen Waasland, Sint-Niklaas
  - Beschut Wonen Veurne-Diksmuide, Veurne

REFERENCES:
- [Derived] Verhaeghe N, Clays E, Vereecken C, De Maeseneer J, Maes L, Van Heeringen C, De Bacquer D, Annemans L. Health promotion in individuals with mental disorders: a cluster preference randomized controlled trial. BMC Public Health. 2013 Jul 15;13:657. doi: 10.1186/1471-2458-13-657. PMID 23855449
- [Derived] Verhaeghe N, De Maeseneer J, Maes L, Van Heeringen C, Bogaert V, Clays E, De Bacquer D, Annemans L. Health promotion intervention in mental health care: design and baseline findings of a cluster preference randomized controlled trial. BMC Public Health. 2012 Jun 13;12:431. doi: 10.1186/1471-2458-12-431. PMID 22694796